CLINICAL TRIAL: NCT06408233
Title: Person-Centered Quality Measurement and Management (QM2) in a System for Addictions Treatment in New York State (Project 3)
Brief Title: Person-Centered Quality Measurement and Management in a System for Addictions Treatment in New York State (Project 3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-00896; 1RM1DA059377-01 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-05-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Health Services Research

STUDY DESIGN:
Intervention Model Description: This study is a stepped wedge design where clinics are randomized to onset of intervention in one of five time periods over the three years of the intervention rollout (years 2-4 of the phase) and tracked using administrative data. Data for all clinic clients during each of the seven six-month periods will be drawn from administrative data. All clinics will be in the control condition for the first six-month period. Seven clinics will be assigned randomly to one of five time periods for onset of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Performance coaching (Experimental): All clinics will receive the performance coaching intervention. There is only one arm to this study.
  Interventions: Other: Performance Coaching

INTERVENTIONS:
Other: Performance Coaching — Performance coaching will consist of working with clinic staff to understand and guide current quality measurement practices as well as improving quality measurement and implementing new measures and management practices.

SUMMARY:
The goal of this study is to implement Opioid Use Disorder Quality Measurement and Management (OUD-QM2) strategy by the Office of Addiction Services and Supports (OASAS) to drive change and improve treatment practices. Through a concurrent mixed methods approach that iteratively examines quantitative and qualitative data to inform the process, the investigators will examine the effects of the strategy on stakeholders-PWUD/patients, families, and providers-and outcomes. This comprehensive approach will allow for a "global" view of the perceived effects of the OUD-QM2 strategy for all stakeholders while allowing us to use administrative data to test the effects of the strategy on patient outcomes. Through qualitative interviews and focus groups conducted in years 1, 3, and 5 of the phase, the investigators will derive information from stakeholders about their perceptions and use of the quality measures. Through surveys conducted with all clinics, the investigators will elicit data on changes in provider use of quality measures, clinical practice, and use of measures for incentive-based contracting. Finally, the investigators will conduct a stepped wedge trial to examine the effects of performance coaching that guides clinics on use of the quality measures for clinical practice improvement. The trial will also benefit from a treatment as usual (TAU) condition of clinics not participating in the trial to examine secular trends in patient outcomes across the period of the OASAS QM2 strategy rollout. The overall aim is to build and test a science-based OUD-QM2 strategy for person-centered treatment.

DETAILED DESCRIPTION:
The NYULH research team in collaboration with OASAS will conduct surveys of all 550 outpatient clinics across the state at three time points, years 1, 3, and 5. The NYULH research team and collaborating sites will observe effects on outcomes for patients in Substance Use Disorder (SUD) treatment clinics using administrative data for all outpatient clinics in the New York OASAS system. The study team will test an organizational-level QM2 intervention by employing a stepped-wedged randomized controlled trial with 35 clinics receiving the performance coaching intervention and the remaining clinics in the system treated as usual (TAU). That is, the study team will be able to track change over time for all clinics throughout the system as well as test the marginal effect of the performance coaching on patient outcomes. The study will test whether the OASAS QM2 strategy increases retention in care and has any effect on adverse events (i.e., emergency department visits, hospitalizations, mortality). Clinics receiving the intervention will be randomized to one of five sequences reflecting different timing of the intervention between years 2 and 4. The examination of outcomes will benefit from access to the rich sources of data described above for phase 1. Qualitative data collection with staff and patients will be embedded within the trial to examine experiences with the intervention and to inform quantitative findings.

NYULH and OASAS will maintain stakeholder engagement throughout the implementation and evaluation of the OASAS OUD-QM2 strategy. The study team will seek input from the stakeholder groups on strategies for presenting quality data as well as providing technical assistance to each group. The stakeholders will also receive annual updates on emerging findings from qualitative interviews and focus groups, surveys, and analyses of administrative data to inform them as well as solicit feedback and support for broader dissemination efforts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age, and older
* Clients and clinicians of people attending substance use treatment programs in New York State with Opioid Use Disorder in the time interval 2020-2027

Exclusion Criteria:

* There are no exclusion criteria related to sex/gender to increase the generalizability of the findings. Children will not be included in this study because the treatment system mostly includes adults.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of substance use related emergency department visits | Baseline (6 months prior to intervention), 6 months post-intervention
Change in number of substance use related hospitalizations | Baseline (6 months prior to intervention), 6 months post-intervention
Change in mortality rate | Baseline (6 months prior to intervention), 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Charles Neighbors, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared but aggregated deidentified data will be available through publications post analysis.